CLINICAL TRIAL: NCT04183127
Title: Exploring Advanced Clinical Practitioner's Experience Developing Clinical Competence and Opinions on Role Identity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Sheffield (Other)
Collaborators: South Yorkshire and Bassetlaw Faculty of Advanced Clinical Practice (Unknown); Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CHC-ACP2019
Record Dates: First submitted 2019-11-22; First posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: ACP; Nurse's Role; Development, Consensus
Keywords: ACP; Competence; Role identity
MeSH Terms: interventions — Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ACP: ACPs, either qualified or in training, working in the South Yorkshire and Bassetlaw area.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — ACPs, qualified or in training, will be invited to participate by email. Interested participants will be provided with study materials and asked to complete an online eligibility questionnaire; if eligible, contact details will also be recorded. Participants will be invited to take part in a focus group about their experience in developing clinical competence and their opinions on role identity. Data collection will consist of focus groups.
  Other Names: Focus Groups

SUMMARY:
In the United Kingdom, there is an urgent need to reshape the National Health Service (NHS) workforce to equip it to meet the changing demands of the population it serves and deliver the vision set out in the Next Steps on the NHS Five Year Forward View (2017) and recently published NHS Plan (2019). One of the key elements to this is the continuing development, support and utilisation of Advanced Clinical Practice (ACP) roles.

Advanced Clinical Practitioners are educated to Masters Level in clinical practice and assessed as competent in practice using their expert clinical knowledge and skills. They have the freedom and authority to act, making their own decisions in the assessment, diagnosis and treatment of patients.

Although the level of education and assessment of competence are common for ACPs working in all areas, training and supervision varies between primary and secondary care, specialties and sites.

The proposed research will explore ACP experiences of how they develop clinical competence and their opinions on role identity, specifically:

* Factors that have influenced their clinical competency achievements.
* Training experience (clinical and external education opportunities)
* Experience of educational/ clinical supervision and its benefits.
* Self-identified knowledge gaps, with a focus on mental health.
* Future ACP role identity

ELIGIBILITY:
Inclusion Criteria:

* Qualified ACP or trainee ACP who has completed at least 1 years (FTE) of ACP clinical training
* Currently working in this role within either Primary or Secondary Care and based in South Yorkshire and Bassetlaw.

Exclusion Criteria:

* Unable to communicate in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants will be NHS staff working in the Yorkshire and Bassetlaw region as ACPs (qualified or in training).
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Experiences and views of ACPs regarding their experience of developing clinical competence and opinions on role identity [Time frame: 120 minutes] | Jan-Dec 2020
  Focus groups will follow a topic guide to explore the factors which influence participants experience of clinical competence, training experience and supervision. The focus groups will also discuss participants feelings in relation to self-identified knowledge gaps (focusing on mental health) and the future ACP role identity.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sheffield, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT04183127/Prot_000.pdf